CLINICAL TRIAL: NCT05912556
Title: Brain Response to an Intervention Using Guided, At-Home Technology for the Mind - A Randomized, Controlled, Double-blinded, Parallel-group Intervention Study to Assess an At-Home Program for Improving Cognition and Inducing Changes in Brain Structure and Function
Brief Title: Brain Response to an Intervention Using Guided, At-Home Technology for the Mind
Acronym: BRIGHT-Mind
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lumos Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LL-015
Record Dates: First submitted 2023-06-08; First posted 2023-06-22 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Cognition; Brain Health; Brain Structure; Brain Function

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Other): Remote-Only subjects
  Interventions: Device: Digital Program 1; Device: Digital Program 2
- Cohort B (Other): Remote + Imaging subjects
  Interventions: Device: Digital Program 1; Device: Digital Program 2

INTERVENTIONS:
Device: Digital Program 1 — 2/3 of randomized subjects use digital program 1 for 12 weeks to provide mental stimulation
Device: Digital Program 2 — 1/3 of randomized subjects use digital program 2 for 12 weeks to provide mental stimulation

SUMMARY:
The objective of this study is to assess the effectiveness of two digital programs for providing mental stimulation, improving cognition, and inducing changes in brain structure and function.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 25-80 years of age.
* Ability to understand and speak English, follow written and verbal instructions (English), and give informed consent (English), as assessed by study staff.
* Ability to comply with all the testing and study requirements, including the ability to independently use a video conferencing tool and the ability to independently use a computer to access the web.
* Ability to independently complete a daily, online intervention and outcome assessments using a web browser compatible with the intervention and assessment software on a reliable, internet-connected laptop or desktop computer.

Exclusion Criteria:

* Current, controlled (requiring treatment) or uncontrolled psychiatric diagnosis, including but not limited to posttraumatic stress disorder, psychosis, bipolar illness, pervasive developmental disorder, severe obsessive compulsive disorder, severe depressive or severe anxiety disorder, conduct disorder, attention-deficit/hyperactivity disorder, or other symptomatic manifestations that in the opinion of the Investigator may confound study data/assessments.
* Current, controlled (requiring treatment) or uncontrolled neurological diagnosis, including but not limited to Alzheimer's Disease, other dementias, mild cognitive impairment, Huntington's Disease, Parkinson's Disease, multiple sclerosis, stroke, epilepsy, aphasia, or other condition that in the opinion of the Investigator may confound study data/assessments.
* Any other medical condition in the last 90 days that in the opinion of the Investigator may confound study data/assessments.
* Has been under the care of a caretaker or has not been living independently in the last 90 days.
* In the last three years has used any of the following for more than two weeks continuously: Online courses, Online brain training programs
* Known sensitivity (such as headaches, dizziness, nausea) to bright, stimulating video displays.
* History of seizures (excluding febrile seizures), or significant motor or vocal tics, including but not limited to Tourette's Disorder and photo-sensitive epilepsy.
* Visual acuity that cannot be corrected that prevents or negatively impacts computer activity.
* Has participated in a clinical trial within 90 days prior to screening.
* Pregnancy or planning to become pregnant.

Additional Exclusion Criteria for Cohort B only:

* Unwillingness or inability to comply with imaging safety protocols.
* Metal implants or exposure to shrapnel.
* Left-handed or ambidextrous.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 816 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2025-03-14 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Overall Composite from Creyos (formerly Cambridge Brain Sciences) | Study Day 0 to Study Day 84
  The Overall Composite is derived from the 12 tests in the Creyos battery.

SECONDARY OUTCOMES:
Concentration Domain Score from Creyos | Study Day 0 to Study Day 84
Memory Domain Score from Creyos | Study Day 0 to Study Day 84
Planning Domain Score from Creyos | Study Day 0 to Study Day 84
Reasoning Domain Score from Creyos | Study Day 0 to Study Day 84
Structural Brain Composite from Magnetic Resonance Imaging (MRI) | Study Day 0 to Study Day 84
White Matter Microstructure Composite from Diffusion Magnetic Resonance Imaging (dMRI) | Study Day 0 to Study Day 84
Within-Network Functional Connectivity from Resting-State functional Magnetic Resonance Imaging (fMRI) | Study Day 0 to Study Day 84

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Madore, PhD, Principal Investigator — Lumos Labs, Inc.
Locations (1):
- Lumos Labs, Inc., San Francisco, California, United States